CLINICAL TRIAL: NCT02968979
Title: Cross-sectional, Multicentric, Non-interventional Study to Assess the Frequency and the Management of Cachexia and Associated Symptoms in Patients With Non-small Cell Lung Cancer.
Brief Title: Non-interventional Study to Assess the Frequency of Cachexia in Patients With Non-small Cell Lung Cancer.
Acronym: CacheMire
Status: Completed | Type: Observational
Sponsor: Chugai Pharma France (Industry)
Collaborators: French College of General Hospital Pneumologists (CPHG) (Other); French-Speaking Association of Supportive Care in Cancer (AFSOS) (Unknown); ITEC Services (Other)
Responsible Party: Sponsor
Other Study IDs: CPF-ANA-001
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Non-small Cell Lung Cancer; Cachexia
Keywords: Cachexia; Non-Small Cell Lung cancer; Anorexia; Malnutrition
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cachexia; Anorexia; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the frequency of cachexia and the management of cachexia and associated symptoms in a patient population with non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is a cross-sectional, non-interventional, European (France and Belgium), multicentric prevalence study, conducted on a representative population of 500 patients with NSCLC, to assess the frequency and the management of cachexia and associated symptoms.

The study will be conducted in accordance with the professional code of ethics and the good epidemiological practices guidelines developed by the ADELF (the Association of French-Speaking Epidemiologists) and in accordance with the STROBE recommendations for the drafting of reports and publications related to the study.

The information will be collected during a single visit to the oncologist/lung specialist as part of the usual patient management of his/her lung cancer. The physician will explain the purpose of the study to the patient with an information form specific to the study and will inform him/her of the option to refuse or withdraw from participation. The patient information form in France or a specific consent form in Belgium will be signed by the patient and a copy will be given to him/her (the original will be kept by the physician).

This study does not require any additional specific data. Data will come from the medical file and from the routine disease management. Furthermore, the following self-completion questionnaires will be proposed to patients: Visual analogue scale for dietary intake (dietary intake VAS), assessment of the concerns associated with the anorexia/cachexia (Anorexia-Cachexia module of the Functional Assessment of Anorexia/Cachexia Therapy [FAACT] questionnaire), quality of life (EORTC QLQ-C30), and assessment of physical activity (IPAQ, International Physical Activity Questionnaire). Abdominal CT-scan, if available, will be collected for assessment of skeletal muscle mass index at L3.

ELIGIBILITY:
Inclusion Criteria:

* Patient 18 years of age and older
* Patient with NSCLC
* Patient who has been informed of the study and who has signed a patient information leaflet for France or an informed consent for Belgium
* Patient able to complete a self-assessment questionnaire

Exclusion Criteria:

* Patient unable to consent and/or unable to sign the patient information form in France or an informed consent in Belgium
* Patient with a complete resection of an early stage NSCLC
* History of head and neck cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with non-small cell lung cancer (NSCLC) from outpatient visit, Day Hospital or in-patient hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 539 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luz Bobadilla, MD, Study Director — Chugai Pharma France
Locations (1):
- Chugai Pharma France, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearon K, Strasser F, Anker SD, Bosaeus I, Bruera E, Fainsinger RL, Jatoi A, Loprinzi C, MacDonald N, Mantovani G, Davis M, Muscaritoli M, Ottery F, Radbruch L, Ravasco P, Walsh D, Wilcock A, Kaasa S, Baracos VE. Definition and classification of cancer cachexia: an international consensus. Lancet Oncol. 2011 May;12(5):489-95. doi: 10.1016/S1470-2045(10)70218-7. Epub 2011 Feb 4. PMID 21296615

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 56 oncologists, lung specialists or radiation oncologists treating patients with a malignant lung tumour have recruited patients from outpatient visit, day hospital or in-patient hospitalization in France and Belgium, between the 25th of July and the 31th of October 2016. Patients were recruited in a consecutive manner.
Pre-assignment Details: 539 patients were recruited. Among them, 5 did not meet the eligibility criteria, 1 withdrew his/her consent, 2 were excluded during the data review because the cancer histology was undefined.
  The analysis population included 531 patients and among them 312 had skeletal muscle mass assessment.
Groups:
- NSCLC Patient: Patients,18 years and older, with Non Small Cell Lung Cancer (NSCLC) regardless of the tumor stage and the treatment line
Period: Overall Study
Arm/Group | NSCLC Patient
Started | 539
Completed | 531 (This cross-sectional study had only 1 visit.)
Not Completed | 8
Not completed — Protocol Violation | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is composed of all included patients without major protocol deviation.
Arm/Group | NSCLC Patient
Number analyzed (Participants) | 531
Age, Continuous [Mean (Standard Deviation); unit: year] | 65.2 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178
  Male | 353
Performance Status ECOG (Eastern Cooperative Oncology Group) [Count of Participants; unit: Participants] — Evaluated by the Investigator during the patient visit (4=worst outcome) :
  0 Fully active - Able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. Capable of only limited self-care. Confined to bed or chair more than 50% of waking hours.
  4. Completely disabled. Cannot carry on any self-care; totally confined to bed or chair.
  Participants
    0 | 124
    1 | 300
    2 | 87
    3 | 19
    4 | 1
Smoking status [Count of Participants; unit: Participants]
  Non smoker | 64
  Past smoker | 359
  Current smoker | 97
  Missing | 11
Histology type [Count of Participants; unit: Participants]
  Squamous cell carcinoma | 140
  Adenocarcinoma | 348
  Large cell carcinoma | 18
  Others | 25
Molecular abnormalities [Count of Participants; unit: Participants] — Population: Missing data for 202 patients
  Participants
    number analyzed (Participants) | 329
    EGFR, ALK, ROS1, BRAF or HER2 | 54
    K-RAS | 61
    None | 214
Tumor stages [Count of Participants; unit: Participants] — TNM stage at the time of the visit was collected by the Investigator and classified as follow:
  * Stage 0: (Tis N0 M0)
  * Stage I - II: (T1a /T1b N0 M0) (T2a N0 M0) (T1a/T1b N1 M0 - T2a N1 M0 - T2b N0 M0) (T2b N1 M0 - T3 N0 M0)
  * Stage III A: (T1/T2 N2 M0 - T3 N1/N2 M0 - T4 N0/N1 M0)
  * Stade III B - IV : (T4 N2 M0 - T1/T2/T3/T4 N3 M0) (T1/T2/T3/T4 N0/N1/N2/N3 M1A/M1 with at least 1 lung/pleura or lymph node metastasis) (T1/T2/T3/T4 N0/N1/N2/N3 M1B/M1 with at least 1 metastasis other than lung/pleura or lymph node metastasis) Population: Missing data for 27 patients
  Participants
    number analyzed (Participants) | 504
    Stage I-II | 34
    Stage IIIA | 21
    Stage IIIB-IV | 440
    Unknown stage | 9

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Cachexia According to Modified Fearon Criteria
Description: Percentage of NSCLC patients with a cachexia according to Fearon criteria modified for the stages of pre-cachexia and refractory cachexia in order to classify all the featured cases without ambiguity.
  A patient was considered to have cachexia if he/she had:
  * Weight loss >5% in the last 6 months prior to inclusion or
  * BMI <20 kg/m² and weight loss between 2 and 5% in the 6 months prior to inclusion or
  * Weight loss >2% and sarcopenia (as evaluated by the muscle mass index at L3) if available. If data were not available regarding possible sarcopenia, the presence of cachexia was assigned based on the 2 above conditions.
  In the 3 cases defined above, patient should not have entered the refractory cachexia stage, which was defined as: ECOG performance score of 3 or 4 and a low survival expectancy as defined by Martin et al. (J Clin Oncol 2015) (BMI <20 kg/m² and weight loss ≥ 6%) or (20 ≤ BMI ≤ 21.9 kg/m² and weight loss ≥ 11%) or (22 kg/m² ≤ BMI and weight loss ≥ 15%).
Time Frame: Day1
Population: missing data for 84 patients
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC Patients With Cachexia: Patients,18 years and older, with Non Small Cell Lung Cancer (NSCLC) regardless of the tumor stage and the treatment line with a cachexia
Arm/Group | NSCLC Patients With Cachexia
Number analyzed (Participants) | 447
Participants | 173

2. Secondary Outcome: Frequency of the Different Stages of Cachexia in the General NSCLC Population
Description: Percentage of the different stages of cachexia at inclusion.
  The different stages of cachexia used the following classification:
  * No Cachexia: 1) no weight loss (WL<2%) or 2) weight gain AND no anorexia AND no sarcopenia
  * The pre-cachexia stage : 1) 2% ≤ weight loss ≤ 5% AND BMI ≥ 20 and/or 2) anorexia (according to question 13 of the quality of life questionnaire QLQ-C30) and/or 3) weight loss < 2% AND sarcopenia
  * Cachexia: 1) Weight loss > 5% OR 2) weight loss between 2 and 5% AND BMI < 20 kg/m² OR 3) weight loss > 2% AND sarcopenia. In all cases, patient should not have entered the refractory cachexia stage
  * Refractory cachexia: ECOG 3 or 4 AND low survival expectancy [BMI < 20kg/m² and weight loss ≥ 6%] OR [20 ≤ BMI ≤ 21,9 kg/m² and weight loss ≥ 11%] OR [22 kg/m² ≤ BMI and weight loss ≥ 15%]
Time Frame: Day 1
Population: Missing data for 84 patients
Measure: Count of Participants; unit: Participants
Groups:
- NSCLC Patients: Patients,18 years and older, with Non Small Cell Lung Cancer (NSCLC) regardless of the tumor stage and the treatment line
Arm/Group | NSCLC Patients
Number analyzed (Participants) | 447
Participants
  No Cachexia | 119
  Pre-Cachexia | 151
  Cachexia | 173
  Refractory Cachexia | 4

3. Secondary Outcome: Frequency of the Different Stages of Cachexia in the General NSCLC Population According to Stage Associated With NSCLC.
Description: Percentage of the different stages of cachexia at inclusion according to the NSCLC stage
Time Frame: Day 1
Population: Patients,18 years and older, with Non Small Cell Lung Cancer (NSCLC) Missing data for 81 patients
Measure: Count of Participants; unit: Participants
Groups:
- Cancer Stage I-II: Patients with one of the following TNMs at the time of the visit: (T1a /T1b N0 M0) (T2a N0 M0) (T1a/T1b N1 M0 - T2a N1 M0 - T2b N0 M0) (T2b N1 M0 - T3 N0 M0)
- Cancer Stage IIIA: Patients with one of the following TNMs at the time of the visit: (T1/T2 N2 M0 - T3 N1/N2 M0 - T4 N0/N1 M0)
- Cancer Stage IIIB- IV: Patients with one of the following TNMs at the time of the visit: (T4 N2 M0 - T1/T2/T3/T4 N3 M0) (T1/T2/T3/T4 N0/N1/N2/N3 M1A/M1 with at least 1 lung/pleura or lymph node metastasis) (T1/T2/T3/T4 N0/N1/N2/N3 M1B/M1 with at least 1 metastasis other than lung/pleura or lymph node metastasis)
Arm/Group | Cancer Stage I-II | Cancer Stage IIIA | Cancer Stage IIIB- IV
Number analyzed (Participants) | 31 | 13 | 370
Participants
  No Cachexia | 9 | 3 | 95
  Pre-Cachexia | 10 | 5 | 124
  Cachexia | 11 | 5 | 148
  Refractory Cachexia | 1 | 0 | 3

4. Secondary Outcome: Frequency of the Different Stages of Cachexia in the General NSCLC Population According to Histology Associated With NSCLC.
Description: Percentage of the different stages of cachexia according to the NSCLC histology
Time Frame: Day 1
Population: Patients,18 years and older, with Non Small Cell Lung Cancer (NSCLC) Missing data for 84 patients
Measure: Count of Participants; unit: Participants
Groups:
- Squamous Cell Carcinoma: Patients with squamous cell carcinoma
- Adenocarcinoma: Patients with adenocarcinoma
- Large Cell Carcinoma and Other Histology Type: Patients with large cell carcinoma and other histology type
Arm/Group | Squamous Cell Carcinoma | Adenocarcinoma | Large Cell Carcinoma and Other Histology Type
Number analyzed (Participants) | 116 | 296 | 35
Participants
  No Cachexia | 35 | 79 | 5
  Pre-Cachexia | 38 | 98 | 15
  Cachexia | 43 | 115 | 15
  Refractory Cachexia | 0 | 4 | 0

5. Secondary Outcome: Frequency of Sarcopenia in the General NSCLC Patients With Cachexia
Description: Percentage of patients with sarcopenia in the general NSCLC patients with cachexia
Time Frame: Day 1
Population: Population with no missing data for the 3 interest criteria defining the cachexia
Measure: Count of Participants; unit: Participants
Groups:
- Cachexia NSCLC Patients: A patient was considered to have cachexia if he/she had:
  * Weight loss >5% in the last 6 months prior to inclusion or
  * BMI <20 kg/m² and weight loss between 2 and 5% in the 6 months prior to inclusion or
  * Weight loss >2% and sarcopenia (as evaluated by the muscle mass index at L3) if available. If data were not available regarding possible sarcopenia, the presence of cachexia was assigned based on the 2 above conditions.
  In the 3 cases defined above, patient should not have entered the refractory cachexia stage, which was defined as: ECOG performance score of 3 or 4 and a low survival expectancy as defined by Martin et al. (J Clin Oncol 2015) (BMI <20 kg/m² and weight loss ≥ 6%) or (20 ≤ BMI ≤ 21.9 kg/m² and weight loss ≥ 11%) or (22 kg/m² ≤ BMI and weight loss ≥ 15%).
Arm/Group | Cachexia NSCLC Patients
Number analyzed (Participants) | 111
Participants | 74

6. Secondary Outcome: Frequency of Sarcopenia With no Clinical Significant Weight Loss in the General NSCLC Patients With Pre-cachexia
Description: Percentage of patient with sarcopenia and no clinical significant weight loss (sarcopenia and WL< 2%) in the general NSCLC patients with pre-cachexia:
Time Frame: Day 1
Population: Population with no missing data for the 3 interest criteria defining the pre-cachexia
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Cachexia NSCLC Patients: Pre-cachexia was defined as:
  * 2% ≤ weight loss (WL) ≤ 5% and BMI ≥ 20 kg/m² or
  * anorexia or
  * sarcopenia and WL< 2%
Arm/Group | Pre-Cachexia NSCLC Patients
Number analyzed (Participants) | 89
Participants | 59

7. Secondary Outcome: Frequency of the Different Stages of Cachexia in the General NSCLC Population According to Molecular Abnormalities Associated With NSCLC.
Description: Percentage of the different stages of cachexia according to the molecular abnormalities associated with NSCLC:
  * EGRF, ALK, ROS1, BRAF or HER2
  * K-RAS
  * No mutation
Time Frame: Day 1
Population: NSCLC patients Overall number of patients analyzed for cachexia stage; 244 missing data.
Measure: Count of Participants; unit: Participants
Groups:
- EGFR, ALK, ROS1, BRAF or HER2: NSCLC patients with at least one of the following molecular abnormalities : EGFR, ALK, ROS1, BRAF or HER2
- K-RAS: NSCLC patients with a K-RAS molecular abnormality
- No Mutation: NSCLC patients with no mutation
Arm/Group | EGFR, ALK, ROS1, BRAF or HER2 | K-RAS | No Mutation
Number analyzed (Participants) | 46 | 58 | 183
Participants
  No Cachexia | 8 | 21 | 48
  Pre-Cachexia | 27 | 13 | 54
  Cachexia | 11 | 24 | 79
  Refractory Cachexia | 0 | 0 | 2
Statistical Analysis 1: Comparison: EGFR, ALK, ROS1, BRAF or HER2 vs K-RAS vs No Mutation; Statistical analysis applies to all rows and columns; Test type: Other; p = 0.0032, likelihood-ratio test
Statistical Analysis 2: Comparison: EGFR, ALK, ROS1, BRAF or HER2 vs K-RAS vs No Mutation; Statistical Analysis 2 for Frequency of the Different Stages of Cachexia, excluding the refractory cachexia stage, in the General NSCLC Population According to Molecular Abnormalities Associated With NSCLC. Statistical analysis applies to all rows and columns; Test type: Other; p = 0.0008, Chi-squared

8. Secondary Outcome: Frequency of the Different Stages of Cachexia According to the Number of Treatments Received.
Description: NSCLC patients. 84 patients with missing data
Time Frame: Day 1
Measure: Count of Participants; unit: Participants
Groups:
- no NSCLC Treatment: Patient with no cancer treatment received for NSCLC
- 1 NSCLC Treatment: Patient with 1 cancer treatment received for NSCLC
- 2 NSCLC Treatments: Patient with 2 cancer treatments received for NSCLC
- 3 NSCLC Treatments: Patient with 3 cancer treatments received for NSCLC
- at Least 4 NSCLC Treatments: Patient with at least 4 cancer treatments received for NSCLC
Arm/Group | no NSCLC Treatment | 1 NSCLC Treatment | 2 NSCLC Treatments | 3 NSCLC Treatments | at Least 4 NSCLC Treatments
Number analyzed (Participants) | 41 | 82 | 137 | 79 | 107
Participants
  No Cachexia | 6 | 18 | 42 | 26 | 27
  Pre-Cachexia | 11 | 31 | 42 | 22 | 44
  Cachexia | 24 | 32 | 50 | 31 | 36
  Refractory Cachexia | 0 | 1 | 3 | 0 | 0

9. Secondary Outcome: Frequency of the Different Stages of Cachexia According to the Types of Treatments Received.
Description: Stage of cachexia at inclusion according to the type of treatments received (surgery, radiotherapy, chemotherapy, targeted therapies).
Time Frame: Day 1
Population: NSCLC patients. 101 missing data
Measure: Count of Participants; unit: Participants
Groups:
- Surgery: Patient who had at least 1 surgery for NSCLC treatment
- Radioterapy: Patient who received at least 1 radiotherapy for NSCLC treatment
- Chemotherapy: Patient who received at least 1 chemotherapy for NSCLC treatment
- Targeted Therapy: Patient with at least 1 targeted therapy received for NSCLC
Arm/Group | Surgery | Radioterapy | Chemotherapy | Targeted Therapy
Number analyzed (Participants) | 39 | 133 | 378 | 79
Participants
  No Cachexia | 7 | 42 | 107 | 16
  Pre-Cachexia | 16 | 50 | 121 | 42
  Cachexia | 16 | 40 | 146 | 21
  Refractory Cachexia | 0 | 1 | 4 | 0

10. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Nutritional State
Description: • Nutritional state according to the different stages of cachexia The variables used will be: serum albumin levels, serum pre-albumin levels, BMI and weight.
Time Frame: Day 1
Population: NSCLC patients
Measure: Count of Participants; unit: Participants
Groups:
- Weight Loss >=15%: Patients with weight loss at inclusion >=15% of the weight 6 months prior to inclusion.
- Weight Loss >=10%: Patients with weight loss at inclusion >=10% of the weight 6 months prior to inclusion.
- Albuminemia < 30-35g/L: Patients with albuminemia < 30g/L (patient < 70 years old) or < 35g/L (patient ≥ 70 years old)
- Pre-albuminemia < 110-200 mg/L: Patients with pre-albuminemia < 110g/L (patient < 70 years old) or < 200 mg/L (patient ≥ 70 years old)
- BMI <18.5-21 kg/m²: BMI at inclusion visit < 18,5 kg/m² (patient < 70 years old) or < 21 kg/m² (patients≥70 years old)
Arm/Group | Weight Loss >=15% | Weight Loss >=10% | Albuminemia < 30-35g/L | Pre-albuminemia < 110-200 mg/L | BMI <18.5-21 kg/m²
Number analyzed (Participants) | 31 | 63 | 35 | 6 | 68
Participants
  No Cachexia | 0 | 0 | 5 | 2 | 8
  Pre-Cachexia | 0 | 0 | 7 | 1 | 20
  Cachexia | 29 | 60 | 21 | 3 | 37
  Refractory Cachexia | 2 | 3 | 2 | 0 | 3

11. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Blood Glucose
Description: Blood glucose abnormalities according to the different stages of cachexia at inclusion
Time Frame: Day 1
Population: NSCLC patients 329 data missing
Measure: Count of Participants; unit: Participants
Groups:
- Normal Blood Glucose: < 1g/L
- Moderate Blood Glucose: >= 1g/L <= 1.26g/L
- High Blood Glucose: >1.26g/L
Arm/Group | Normal Blood Glucose | Moderate Blood Glucose | High Blood Glucose
Number analyzed (Participants) | 56 | 36 | 26
Participants
  No cachexia | 14 | 5 | 4
  Pre-cachexia | 20 | 15 | 12
  Cachexia | 21 | 16 | 10
  Refractory cachexia | 1 | 0 | 0

12. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Loss of Appetite - Dietary Intake Visual Analog Scale
Description: Dietary Intake Visual Analog Scale (Dietary intake VAS): The question "Could you indicate the amount you currently eat, placing a vertical mark on the line between "nothing at all" and "as usual"? ". Depending on the location of the patient mark on the scale, a score of between 0 ("nothing at all") and 10 ("as usual") will be allocated.
Time Frame: Day 1
Population: NSCLC patients 12 missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- No Cachexia: 1) no weight loss (WL<2%) or 2) weight gain AND no anorexia AND no sarcopenia
- Pre-cachexia: 1) 2% ≤ weight loss ≤ 5% AND BMI ≥ 20 and/or 2) anorexia (according to question 13 of the quality of life questionnaire QLQ-C30) and/or 3) weight loss < 2% AND sarcopenia
- Cachexia: 1) Weight loss > 5% OR 2) weight loss between 2 and 5% AND BMI < 20 kg/m² OR 3) weight loss > 2% AND sarcopenia. In all cases, patient should not have entered the refractory cachexia stage
- Refractory Cachexia: ECOG 3 or 4 AND low survival expectancy [BMI < 20kg/m² and weight loss ≥ 6%] OR [20 ≤ BMI ≤ 21,9 kg/m² and weight loss ≥ 11%] OR [22 kg/m² ≤ BMI and weight loss ≥ 15%]
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 117 | 146 | 168 | 4
score on a scale | 9.57 (1.07) | 7.68 (2.64) | 6.51 (2.89) | 3.13 (1.16)

13. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Loss of Appetite - AC/S FAACT
Description: Score of the 12-question AC/S module (Anorexia-Cachexia module) of the Functional Assessment of Anorexia/Cachexia Therapy (FAACT) questionnaire assessing anorexia and cachexia: the AC/S module of the FAACT questionnaire consists of 12 questions to assess over the last 7 days quality of life, related to anorexia or cachexia. The score ranges between 0 and 48, the higher the score, the higher the quality of life.
Time Frame: Day 1
Population: NSCLC patients 9 missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 119 | 148 | 167 | 4
score on a scale | 40.00 (3.90) | 35.09 (7.02) | 32.60 (7.16) | 25.75 (10.05)

14. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Inflammation Markers - Neutrophil/Lymphocyte Ratio
Description: neutrophil/lymphocyte ratio
Time Frame: Day 1
Population: NSCLC patients 112 missing data
Measure: Median (Inter-Quartile Range); unit: no unit (ratio)
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 86 | 113 | 132 | 4
no unit (ratio) | 2.54 [1.90 to 3.87] | 2.73 [1.85 to 4.37] | 3.75 [2.00 to 6.14] | 7.15 [3.51 to 15.27]

15. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Inflammation Markers - CRP
Description: CRP level
Time Frame: Day 1
Population: NSCLC patients 317 missing data
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 27 | 37 | 64 | 2
mg/L | 18 [5.60 to 30.10] | 7 [3.00 to 25.00] | 21.5 [7.85 to 53.00] | 16.5 [15.00 to 18.00]

16. Secondary Outcome: Description of the Clinical Signs/Symptoms Associated With the Different Stages of Cachexia: Inflammation Markers - Fibrinogen
Description: fibrinogen level
Time Frame: Day 1
Population: NSCLC patients 387 missing data
Measure: Median (Inter-Quartile Range); unit: g/L
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 17 | 18 | 25 | 0
g/L | 4.58 [3.93 to 5.30] | 4.75 [3.90 to 5.90] | 4.96 [4.50 to 6.50] |

17. Secondary Outcome: Description of the Quality of Life Associated With the Different Stages of Cachexia.
Description: Quality of life has been analysed using scores from the functional scale of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire- Core 30 items (EORTC QLQ-C30 questionnaire): score ranging from 0 (malfunction) to 100 (healthy level of functioning) for the following parameters : physical, role, cognitive, emotional and social scales
Time Frame: Day 1
Population: NSCLC patients Physical scale: 16 missing data Role scale: 17 missing data Cognitive scale: 16 missing data Emotional scale: 16 missing data Social scale: 18 missing data
Measure: Mean (Standard Deviation); unit: Scale score
Groups:
- Physical Scale; Role Scale; Cognitive Scale; Emotional Scale; Social Scale: score ranging from 0 (malfunction) to 100 (healthy level of functioning)
Arm/Group | Physical Scale | Role Scale | Cognitive Scale | Emotional Scale | Social Scale
Number analyzed (Participants) | 431 | 430 | 431 | 431 | 429
Scale score
  No Cachexia: number analyzed (Participants) | 119 | 119 | 118 | 118 | 118
  No Cachexia | 76.6 (20.1) | 77.6 (26.9) | 84.5 (21.0) | 82.0 (18.2) | 84.9 (21.3)
  Pre-Cachexia: number analyzed (Participants) | 146 | 146 | 145 | 145 | 144
  Pre-Cachexia | 67.0 (21.4) | 62.6 (32.5) | 79.7 (23.4) | 71.5 (25.1) | 72.0 (28.9)
  Cachexia: number analyzed (Participants) | 162 | 161 | 164 | 164 | 163
  Cachexia | 62.8 (24.5) | 56.2 (35.5) | 79.1 (22.3) | 68.1 (24.8) | 67.8 (31.7)
  Refractory Cachexia: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4
  Refractory Cachexia | 13.3 (9.4) | 0.0 (0.0) | 83.3 (19.2) | 45.8 (35.0) | 12.5 (8.3)
Statistical Analysis 1: Comparison: Physical Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 2: Comparison: Physical Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis — Without refractory cachexia; Without refractory cachexia
Statistical Analysis 3: Comparison: Role Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 4: Comparison: Role Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis — Without refractory cachexia; Without refractory cachexia
Statistical Analysis 5: Comparison: Cognitive Scale; Statistical analysis compares all cachexia stages; Test type: Other; p = 0.1085, Kruskal-Wallis
Statistical Analysis 6: Comparison: Cognitive Scale; Statistical analysis compares all cachexia stages; Test type: Other; p = 0.0482, Kruskal-Wallis — Without refractory cachexia; Without refractory cachexia
Statistical Analysis 7: Comparison: Emotional Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 8: Comparison: Emotional Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis — Without refractory cachexia; Without refractory cachexia
Statistical Analysis 9: Comparison: Social Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis
Statistical Analysis 10: Comparison: Social Scale; Statistical analysis compares all cachexia stages; Test type: Other; p < 0.0001, Kruskal-Wallis — Without refractory cachexia; Without refractory cachexia

18. Secondary Outcome: Description of the Level of Physical Activity Associated With the Different Stages of Cachexia.
Description: Three levels of physical activity are defined:
  1. - Low
     * No activity is reported OR
     * An activity is reported but does not reach moderate or high levels.
  2. - Moderate
     Corresponds to one of the following 3 criteria:
     * 3 or more days of intense activity lasting at least 20 min per day OR
     * 5 or more days of moderate intensity activity and / or walking for at least 30 min per day OR
     * 5 or more days of activity combining walking, activities of moderate or high intensity, thus achieving at least 600 MET-minutes / week
  3. - High
  Corresponds to one of the following 2 criteria:
  * Intense activity at least 3 days a week and at least 1500 MET-minutes / week OR
  * 7 or more days of activity combining walking, moderate and high intensity activities, achieving at least 3000 MET-minutes / week
Time Frame: Day 1
Population: NSCLC patients 69 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 102 | 128 | 144 | 4
Participants
  Low | 30 | 56 | 78 | 4
  Moderate | 34 | 42 | 39 | 0
  High | 38 | 30 | 27 | 0

19. Secondary Outcome: Number of Participants Receiving a Pharmacological Treatment for Cachexia or for Associated Symptoms
Description: Pharmacological treatment of cachexia or associated symptoms: Yes / No
Time Frame: Day 1
Population: NSCLC patients 225 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 47 | 69 | 103 | 3
Participants | 0 | 0 | 1 | 0

20. Secondary Outcome: Number of Participants Receiving a Non-Pharmacological Treatment for Cachexia or for Associated Symptoms
Description: Non-pharmacological treatment of cachexia or associated symptoms: Y/N
Time Frame: Day 1
Population: NLSCS patients with a nutritional consultation within 2 months before inclusion
  1 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 25 | 42 | 80 | 3
Participants | 24 | 41 | 77 | 3

21. Secondary Outcome: Number of Participants Receiving Systemic Corticosteroids, Anti-inflammatory Drugs, Omega 3 Fatty Acids Treatments
Description: Treatments with systemic corticosteroids, anti-inflammatory drugs, Omega 3 fatty acids: Yes/No
Time Frame: Day 1
Population: NSCLC patients 11 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 118 | 148 | 166 | 4
Participants | 35 | 60 | 76 | 3

22. Secondary Outcome: Number of Participants With Diabetes Treatments
Description: Diabetes treatments : Yes/No
Time Frame: Day 1
Population: NSCLC patients 6 missing data
Measure: Count of Participants; unit: Participants
Arm/Group | No Cachexia | Pre-cachexia | Cachexia | Refractory Cachexia
Number analyzed (Participants) | 117 | 151 | 169 | 4
Participants | 9 | 15 | 20 | 0

23. Secondary Outcome: Comparison of the Proportion of Patients With Cachexia, Anorexia and Malnutrition According to the Subjective Assessment of the Clinician and the Different Objective Assessment Criteria: Cachexia
Description: * Proportion of patients with cachexia according to the subjective assessment of the clinician
  * Proportion of patients with cachexia according to the Fearon criteria
Time Frame: Day 1
Population: NSCLC patients Cachexia according to Investigator: 4 missing data Cachexia according to Fearon criteria: 84 missing data
Measure: Count of Participants; unit: Participants
Groups:
- Cachexia According to Investigator: Patients with cachexia according to the subjective assessment of the clinician
- Cachexia According to Fearon Criteria: 1) Weight loss > 5% OR 2) weight loss between 2 and 5% AND BMI < 20 kg/m² OR 3) weight loss > 2% AND sarcopenia. In all cases, patient should not have entered the refractory cachexia stage
Arm/Group | Cachexia According to Investigator | Cachexia According to Fearon Criteria
Number analyzed (Participants) | 527 | 447
Participants | 53 | 173

24. Secondary Outcome: Comparison of the Proportion of Patients With Cachexia, Anorexia and Malnutrition According to the Subjective Assessment of the Clinician and the Different Objective Assessment Criteria: Anorexia
Description: * Proportion of patients with anorexia according to the subjective assessment of the clinician
  * Proportion of patients with anorexia according to the Ingesta VAS
  * Proportion of patients with anorexia according to the AC/S-FAACT module score
  * Proportion of patients with anorexia according to question 13 of the QLQ-C30 questionnaire: "Have you had a lack of appetite?"
Time Frame: Day 1
Population: NSCLC patients Anorexia according to Investigator: 3 missing data Anorexia according to VAS: 22 missing data Anorexia according to FAACT: 19 missing data Anorexia according to question 13 of QLQ-C30 questionnaire: 33 missing data
Measure: Count of Participants; unit: Participants
Groups:
- Anorexia According to Investigator: Patients with anorexia according to the subjective assessment of the clinician
- Anorexia According to VAS: Patients with anorexia according to Visual analogue scale for dietary intake.: "Could you indicate the amount you currently eat, placing a vertical mark on the line between "nothing at all" and "as usual"? Depending on the location of the patient mark on the scale, a score of between 0 ("nothing at all") and 10 ("as usual") was allocated.
  anorexia if score*100/990< 70mm.
- Anorexia According to FAACT: Patients with anorexia according to Anorexia Cachexia/Subcale (AC/S) module of the Functional Assessment of Anorexia/Cachexia Treatment (FAACT) questionnaire: anorexia if score <=37
- Anorexia According to Question 13 of QLQ-C30 Questionnaire: Patients with anorexia according to question 13 of the QLQ-C30 questionnaire: "Have you had a lack of appetite?": anorexia if answer is a A little bit, Somewhat, Quite a bit
Arm/Group | Anorexia According to Investigator | Anorexia According to VAS | Anorexia According to FAACT | Anorexia According to Question 13 of QLQ-C30 Questionnaire
Number analyzed (Participants) | 528 | 509 | 512 | 498
Participants | 109 | 166 | 273 | 219

25. Secondary Outcome: Comparison of the Proportion of Patients With Cachexia, Anorexia and Malnutrition According to the Subjective Assessment of the Clinician and the Different Objective Assessment Criteria: Malnutrition
Description: * Proportion of patients with severe malnutrition according to the subjective assessment of the clinician
  * Proportion of patients with severe malnutrition according to the malnutrition criteria defined by the HAS.
Time Frame: Day 1
Population: NSCLC patients Severe malnutrition according to Investigator: 15 missing data Severe malnutrition according to the HAS: 416 missing data
Measure: Count of Participants; unit: Participants
Groups:
- Severe Malnutrition According to Investigator: Patients with severe malnutrition according to the subjective assessment of the clinician
- Severe Malnutrition According to the HAS: Patients with malnutrition according to the Haute Autorité de Santé:
  * weight loss ≥ 10%,
  * BMI measured during the inclusion visit <18.5 kg / m² for patients aged 70 and under and <21 kg / m² for patients over 70 years of age
  * Albumin <30 g / L if patient <70 years; or albumin <35g / L if patient ≥ 70 years
  * Pre-albumin <110 mg / L if patient <70 years
Arm/Group | Severe Malnutrition According to Investigator | Severe Malnutrition According to the HAS
Number analyzed (Participants) | 516 | 115
Participants | 52 | 55

ADVERSE EVENTS:
Description: This is a non-interventional epidemiological study. No safety data was collected. No reporting of adverse reaction is expected in the study.
Groups:
- No Safety Data Was Collected: This is a non-interventional epidemiological study. No reporting of adverse reaction is expected in the study.
Arm/Group | No Safety Data Was Collected
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study may not be published by the Health Institution or the Investigator without the prior written consent of the Promoter who has to respond as soon as possible.

If the Investigator wishes to proceed with a publication or communication relating to the Study, the Promoter may, in the event that a serious and valid reason appears to require it, request that certain modifications be made. The modifications cannot in any way affect the scientific value of the publication.